CLINICAL TRIAL: NCT02303847
Title: Ultra-low Dose Oral Ketamine for Treatment of Chronic Non-cancer Pain in the Primary Care Setting
Brief Title: Ultra-low Dose Oral Ketamine for Chronic Pain in the Primary Care Setting
Acronym: Ketamine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lucinda Grande, Primary Care Physician, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20141809
Record Dates: First submitted 2014-11-25; First posted 2014-12-01 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Drug (Active Comparator): ketamine 16 mg in flavored syrup by mouth twice daily for 1 week, then ketaming 32 mg in flavored syrup by mouth twice daily for 1 week
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Flavored syrup (without ketamine) by mouth twice daily for 2 weeks

INTERVENTIONS:
Drug: Ketamine — ultra-low dose oral ketamine twice daily in two different doses over a 2 week period.
  Arms: Active Drug

SUMMARY:
This project is a pilot study to evaluate the analgesic and opioid-sparing effects of ketamine in an ultra-low dose oral formulation as a novel intervention for treatment of chronic non-cancer pain in opioid-tolerant patients in the primary care outpatient setting.

DETAILED DESCRIPTION:
Chronic pain is a major national public health issue, affecting about 100 million adults in the United States. Opioid pain medications are commonly used for treatment of chronic pain, but their use is fraught with consequences including an increasing prevalence of misuse, abuse, and overdose death, and side effects which lead to a reduced quality of life. An effective and safe medication that would improve control of chronic pain while reducing reliance on opioid medications would be valuable for patients, medical providers and society at large.

Ketamine, commonly used as an intravenous anesthetic agent, has been shown to have analgesic and opioid-sparing effects in the peri-operative period and in the palliative care setting. Based on promising preliminary data from an open-label treatment trial, this project is a pilot study to evaluate the analgesic and opioid-sparing effects of ketamine in an ultra-low dose oral formulation as a novel intervention for treatment of chronic non-cancer pain in the primary care outpatient setting.

The design of the proposed study is a randomized controlled two week parallel-group trial, with 32 patients receiving either the active treatment or placebo twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Routine use of an opioid medication for non-cancer pain for more than six months
* A current average daily dose of greater than or equal to 20 mg morphine or equivalent
* Current prescription of an as-needed opioid suitable for downward titration during the study period
* Ability to provide informed consent Ability to adhere to the study protocol

Exclusion Criteria:

* Uncontrolled hypertension, cardiac arrhythmia or other known cardiac disease,
* elevated intracranial pressure,
* severe glaucoma,
* schizophrenia,
* diagnosed substance use disorder, or
* other unstable medical or psychiatric illness or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Pain improvement (Brief Pain Inventory (BPI) Mean Pain Severity Scale) | 2 weeks
  Improvement after 2 weeks in pain as measured by the Brief Pain Inventory (BPI) Mean Pain Severity Scale
Function improvement (BPI Mean Interference Scale) | 2 weeks
  Improvement after 2 weeks in functional status as measured by the BPI Mean Interference Scale

SECONDARY OUTCOMES:
Reduction in opioid use (self-reported average opioid dose) | 2 weeks
  Reduction after two weeks in self-reported average opioid dose, converted to morphine equivalents.

OTHER OUTCOMES:
Reduction in depression (PHQ-9 depression score) | 2 weeks
  Reduction in depression, using the PHQ-9 depression score

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Grande, MD, Principal Investigator — University of Washington Department of Family Medicine
Locations (1):
- Pioneer Family Practice, Lacey, Washington, United States